CLINICAL TRIAL: NCT04656535
Title: A Multi-Center Phase 0/I Trial of Anti-TIGIT Antibody AB154 in Combination With Anti-PD-1 Antibody AB122 for Recurrent Glioblastoma.
Brief Title: AB154 Combined With AB122 for Recurrent Glioblastoma
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Arcus Biosciences, Inc. (Industry)
Responsible Party: Principal Investigator, Sylvia Kurz, Associate Professor of Neurology, Yale University
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: 2000028799; R01CA266757 (NIH)
Record Dates: First submitted 2020-11-18; First posted 2020-12-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Glioblastoma
Keywords: Glioblastoma; Recurrent; PD1; TIGIT; Immunotherapy
MeSH Terms: conditions — Glioblastoma; Recurrence | interventions — zimberelimab

STUDY DESIGN:
Intervention Model Description: After the initial safety cohort confirms the safety of the dosing schedule an expansion surgical cohort will be enrolled and this cohort will be randomized to one of four treatment arms for the first cycle prior to surgery,
Who Masked: Participant, Care Provider, Investigator
Masking Description: Masking will only occur in the surgical cohort B (4 arms) during the first cycle prior to surgery. The masking will be removed after surgery and all patients will receive open label treatment with both zimberelimab and domvanalimab.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Zimberelimab (AB 122) + Domvanalimab (AB 154) Safety Cohort (Cohort A) (Experimental): Eligible patients will be sequentially enrolled to receive intravenous domvanalimab (AB 154) combined with zimberelimab (AB 122) (N=6). domvanalimab (AB 154) will be given at a dose of 10 mg/kg and zimberelimab (AB 122) will be given at a dose of 240 mg (flat).
  Interventions: Drug: Zimberelimab; Drug: Domvanalimab
- Domvanalimab (AB 154) Surgical Cohort (Cohort B1) (Experimental): Candidates for surgical resection will be enrolled and initiate study treatment approximately two weeks prior to the resection. The pre-surgical dose (neoadjuvant treatment) will be double-blinded.
  B1 (N=10): domvanalimab (AB 154) single agent (10 mg/kg) + placebo
  Following surgery, all patients will initiate treatment with the combination of domvanalimab (AB 154) and zimberelimab (AB 122). Domvanalimab (AB 154) will be given at a dose of 10 mg/kg and zimberelimab (AB 122) will be given at a dose of 240 mg (flat).
  Interventions: Drug: Domvanalimab; Drug: Placebo
- Zimberelimab (AB 122) Surgical Cohort (Cohort B2) (Experimental): Candidates for surgical resection will be enrolled and initiate study treatment approximately two weeks prior to the resection. The pre-surgical dose (neoadjuvant treatment) will be double-blinded.
  B2 (N=10): zimberelimab (AB 122) single agent (240 mg) + placebo
  Following surgery, all patients will initiate treatment with the combination of domvanalimab (AB 154) and zimberelimab (AB 122). Domvanalimab (AB 154) will be given at a dose of 10 mg/kg and zimberelimab (AB 122) will be given at a dose of 240 mg (flat).
  Interventions: Drug: Zimberelimab; Drug: Placebo
- Domvanalimab (AB 154) + Zimberelimab (AB 122) Surgical Cohort (Cohort B3) (Experimental): Candidates for surgical resection will be enrolled and initiate study treatment approximately two weeks prior to the resection. The pre-surgical dose (neoadjuvant treatment) will be double-blinded.
  B3 (N=10): domvanalimab (AB 154, 10 mg/kg) + zimberelimab (AB 122, 240 mg)
  Following surgery, all patients will initiate treatment with the combination of domvanalimab (AB 154) and zimberelimab (AB 122). Domvanalimab (AB 154) will be given at a dose of 10 mg/kg and zimberelimab (AB 122) will be given at a dose of 240 mg (flat).
  Interventions: Drug: Zimberelimab; Drug: Domvanalimab
- Placebo Surgical Cohort (Cohort B4) (Experimental): Candidates for surgical resection will be enrolled and initiate study treatment approximately two weeks prior to the resection. The pre-surgical dose (neoadjuvant treatment) will be double-blinded.
  B4 (N=10): Two placebo infusions
  Following surgery, all patients will initiate treatment with the combination of domvanalimab (AB 154) and zimberelimab (AB 122). Domvanalimab (AB 154) will be given at a dose of 10 mg/kg and zimberelimab (AB 122) will be given at a dose of 240 mg (flat).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Zimberelimab — Zimberelimab (AB122) is a fully human immunoglobulin G4 (hIgG4) monoclonal antibody (mAb) that targets PD-1.
  Arms: Domvanalimab (AB 154) + Zimberelimab (AB 122) Surgical Cohort (Cohort B3); Zimberelimab (AB 122) + Domvanalimab (AB 154) Safety Cohort (Cohort A); Zimberelimab (AB 122) Surgical Cohort (Cohort B2)
Drug: Domvanalimab — Domvanalimab (AB 154) is a humanized immunoglobulin G1 (IgG1) monoclonal antibody that targets TIGIT.
  Arms: Domvanalimab (AB 154) + Zimberelimab (AB 122) Surgical Cohort (Cohort B3); Domvanalimab (AB 154) Surgical Cohort (Cohort B1); Zimberelimab (AB 122) + Domvanalimab (AB 154) Safety Cohort (Cohort A)
Drug: Placebo — Saline placebo comparator for pre-surgery treatment in cohort B4
  Arms: Domvanalimab (AB 154) Surgical Cohort (Cohort B1); Placebo Surgical Cohort (Cohort B4); Zimberelimab (AB 122) Surgical Cohort (Cohort B2)

SUMMARY:
This is a phase 0/I exploratory study. Patients at first or second recurrence of glioblastoma will be enrolled. The study will be divided into two cohorts: Cohort A (safety cohort) and Cohort B (surgical patient cohort).

Cohort A: Eligible patients will be sequentially enrolled to receive intravenous domvanalimab combined with zimberelimab (N=6). Domvanalimab will be given at a dose of 10 mg/kg and zimberelimab will be given at a dose of 240 mg (flat). The dosing was determined in a separate study in solid tumors; this cohort will confirm the safety of the dosing schedule in patients with brain tumors.

Cohort B: Expansion surgical cohort. The purpose of cohort B is to provide an additional safety evaluation of domvanalimab + zimberelimab as well as tissue and blood for exploratory ancillary studies investigating the effects of domvanalimab + zimberelimab in the tumor and tumor microenvironment. A total of 46 patients will be enrolled in this cohort.

DETAILED DESCRIPTION:
This is a phase 0/I exploratory study. Patients at first or second recurrence of glioblastoma will be enrolled. The study will be divided into two cohorts: Cohort A (safety cohort) and Cohort B (surgical patient cohort).

Cohort A: Eligible patients will be sequentially enrolled to receive intravenous domvanalimab combined with zimberelimab (N=6). Domvanalimab will be given at a dose of 10 mg/kg and zimberelimab will be given at a dose of 240 mg (flat). The dosing was determined in a separate study in solid tumors; this cohort will confirm the safety of the dosing schedule in patients with brain tumors.

Cohort B: Expansion surgical cohort. The purpose of cohort B is to provide an additional safety evaluation of domvanalimab + zimberelimab as well as tissue and blood for exploratory ancillary studies investigating the effects of domvanalimab + zimberelimab in the tumor and tumor microenvironment. A total of 46 patients will be enrolled in this cohort.

Following completion of cohort A, patients who are candidates for surgical resection for management of tumor progression (i.e. need for diagnostic confirmation or tumor debulking) will be enrolled prior to surgical resection, and initiate study treatment approximately two weeks prior to the resection.

Patients will be randomized to one of the four treatment arms and initiate treatment prior to surgery, according to treatment assignment.

The pre-surgical dose (neoadjuvant treatment) will be double-blinded, to minimize dropouts. A total of 10 patients will be allocated to each one of the following groups in a blinded fashion, approximately two weeks before surgery:

* B1 (N=10): domvanalimab single agent (10 mg/kg) + placebo
* B2 (N=10): zimberelimab single agent (240 mg) + placebo
* B3 (N=10): domvanalimab (10 mg/kg) +zimberelimab (240 mg)
* B4 (N=10): Two placebo infusions

Two to six weeks, following surgery, all patients (N=46) will be re-screened and if still eligible will initiate treatment with the combination of domvanalimab and zimberelimab.

ELIGIBILITY:
Inclusion Criteria:

1. Grade IV glioma (glioblastoma and its variants according to the World Health Organization 2021), confirmed in tissue at time of initial diagnosis. Tumors with an IDH 1 or 2 mutation are excluded. Sequencing of IDH 1 and 2 is not required but, at a minimum, a negative result for the presence of IDH-1 R132H mutation on IHC is required for eligibility.
2. First or second recurrence after treatment. Prior treatment must include at least radiation therapy.
3. Measurable contrast enhancing tumor by Response Assessment in Neuro-Oncology (RANO) criteria. Not required for post-surgery eligibility for treatment in cohort B.
4. Age ≥18 years.
5. Karnofsky performance status ≥80 (≥ 70 for eligibility for treatment after surgery in cohort B).
6. Patients must have adequate organ and marrow function as defined below within 14 days of treatment

   * Absolute neutrophil count (ANC) ≥1,500 /mcL
   * Platelets ≥100,000 / mcL
   * Hemoglobin ≥9 g/dL or ≥ 5.6 mmol/L without transfusion or Erythropoietin (EPO) dependency (within 7 days of assessment)
   * Serum creatinine ≤1.5 X upper limit of normal (ULN) OR measured or calculated creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≥ 60 mL/min for subject with creatinine levels > 1.5 X institutional ULN
   * Serum total bilirubin ≤ 1.5 X ULN OR direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN
   * aspartate aminotransferase (SGOT) and alanine transaminase (SGPT) ≤ 2.5 X ULN
   * Albumin >2.5 mg/dL
   * International Normalized Ratio (INR) or Prothrombin Time (PT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
   * Activated Partial Thromboplastin Time (aPTT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
7. An interval of >=12 weeks from the end of prior radiation therapy is required unless there is either: i) histopathologic confirmation of recurrent tumor, or ii) new enhancement on MRI outside of the radiation treatment field.
8. An interval of >=4 weeks or 5 half-lives (whichever is shorter) after the last administration of any investigational agent or any other treatment prior to first study dose.
9. Female subjects of childbearing potential should have a negative urine or serum pregnancy test. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. Female subjects of childbearing potential must be willing to use 2 methods of birth control or be surgically sterile or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year. Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.
10. Ability to understand and the willingness to sign a written informed consent document.

    ADDITIONAL CRITERIA FOR COHORT B
11. Deemed a candidate for tumor debulking, as determined by the neurosurgeon.

Exclusion Criteria:

1. Patients who have been treated with bevacizumab. Note: Previous use of intra-arterial bevacizumab may be allowed, contingent upon review and approval by study principal investigator and sponsor.
2. Patients who have not recovered from adverse events due to prior therapy (i.e. >Grade 1) with the exception of alopecia and fatigue.
3. Patients with multifocal disease. (Cohort B only)
4. Subjects requiring escalating or chronic supraphysiologic doses of corticosteroids (> 10 mg/d of prednisone equivalent or > 2 mg dexamethasone) for control of disease at the time of registration.
5. Patients receiving previous or current treatment with an immune checkpoint inhibitor.
6. Patients with a known diagnosis of immunodeficiency, including Human Immunodeficiency Virus (HIV) or acquired immunodeficiency syndrome (AIDS).
7. Has known active Hepatitis B (e.g., Hepatitis B surface antigen reactive) or Hepatitis C (e.g., Hepatitis C Virus RNA [qualitative] is detected)
8. Has a known history of active tuberculosis (Bacillus Tuberculosis).
9. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
10. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
11. Has known history of, or any evidence of active, non-infectious pneumonitis.
12. Has an active infection requiring systemic therapy.
13. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
14. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
15. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
16. Unable to undergo MRI of the brain with and without contrast enhancement (i.e. pacemaker, allergy to MRI contrast agent or any other contraindication for MRIs).
17. Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2021-04-21 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] associated with the combination AB122 and AB154 in patients with recurrent glioblastoma | through study completion, an average of 2 years
  Adverse events will be listed individually by patient and treatment group. The number of patients experiencing each adverse event will be summarized by organ and grade. The number and percentage of patients with adverse events in the different categories will be summarized by treatment group.

SECONDARY OUTCOMES:
Single cell RNA sequencing of tumor and blood after exposure to AB154 with and without AB122 | through study completion, an average of 2 years
  Pharmacodynamic effects of each pre-surgery treatment will be evaluated with single-cell RNA sequencing of tumor and blood to determine effects of each intervention on the immune response.
Tregs and CD8 T cells ratio by immunofluorescence | through study completion, an average of 2 years
  Resected tumors in cohorts B1 to 4 will be analyzed utilizing immunofluorescence for the ratio between Tregs and CD8 T cells, calculated by counting cells that are positive for a FoxP3 or a CD8 staining.

CONTACTS AND LOCATIONS:
Overall Officials: Sylvia Kurz, MD, Principal Investigator — Professor of Neurology
Locations (3):
- United States (3):
  - University of California San Francisco, San Francisco, California
  - Yale University, New Haven, Connecticut
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No